CLINICAL TRIAL: NCT04785729
Title: To Evaluate the Safety and Efficacy of Almonertinib Combined With Pyrotinib in the Treatment of Advanced NSCLC Patients With HER-2 Amplification/Mutation After EGFR-TKI Resistance: a Multicenter, Open-label Trial
Brief Title: Almonertinib Combined With Pyrotinib in the Treatment of Advanced NSCLC Patients With HER-2 Amplification/Mutation After EGFR-TKI Resistance
Acronym: APPEAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: YX-L-202009/MA-NSCLC-II-014
Record Dates: First submitted 2021-01-25; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- almonertinib (Experimental)
  Interventions: Drug: Almonertinib combine with Pyrrolitinib

INTERVENTIONS:
Drug: Almonertinib combine with Pyrrolitinib — 110mg,qd Almonertinib+（240mg/320mg/400mg）,qd Pyrrolitinib

SUMMARY:
This is a multicenter, open, phase II clinical trial to evaluate the safety and efficacy of almonertinib combined with pyrrolitinib in locally advanced or metastatic NSCLC patients with her-2 variants detected after first-line EGFR-TKI treatment resistance. Patients with first-line EGFR-TKI resistance showed HER-2 variation (including mutation and amplification) in tissue or blood tests, and the treatment regimen of metinil combined with pyrrolitinib was performed to evaluate the safety and efficacy of the treatment regimen. To determine the optimal dose of pyrrolitinib, three dose groups of 240mg, 320mg, and 400mg were set, and the "3+3" study design principle was adopted. About 27-36 people will be included in the study (depending on the progress of the study)

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 ≤ age ≤75, regardless of gender. 2. Non-squamous NSCLC (including stage IIIB-IV patients who relapsed after previous surgical treatment or were newly diagnosed). According to AJCC edition 8 lung cancer Staging Criteria) 3. Previous treatment with EGFR-TKI (not limited to algebra) and radiographic disease progression were permitted with less than or equal to first-line chemotherapy.

  4. Before inclusion in this study (after the last treatment), tumor tissues or blood samples were detected with EGFR-sensitive 19 exon deletion or L858R mutation (with or without T790M), and her-2 mutation (including sensitive mutation or amplification, in which amplification should be confirmed by FISH).

  5. The Eastern Tumor Tissue Cooperative Group (ECOG) physical status score was 0 or 1 and did not deteriorate in the previous 2 weeks, with a minimum expected survival of 12 weeks.

  6. The patient had at least one tumor lesion that had not received previous local treatment such as irradiation, nor had he received biopsy during the screening period, and it could be accurately measured at baseline, with the longest diameter ≥ 10mm at baseline (short diameter ≥ 15mm for lymph nodes). The measurement method chosen is suitable for accurate repeated measurements and can be computed tomography (CT) or magnetic resonance imaging (MRI). If there is only one measurable lesion and no previous local treatment such as irradiation, it may be accepted as the target lesion, and a baseline evaluation of the tumor lesion shall be conducted at least 14 days after the diagnostic biopsy.

  7. For fertile women, appropriate contraception should be used and breastfeeding should not be performed for 3 months from screening to discontinuation of study treatment. A pregnancy test is negative before administration, or there is no proven risk of pregnancy if one of the following criteria is met: A. Postmenopause is defined as amenorrhea over the age of 50 and at least 12 months after cessation of all exogenous hormone replacement therapy.

B. Women younger than 50 years of age may also be considered postmenopausal if they stop all exogenous hormone therapy for 12 months or more and their luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within the laboratory post-menopausal reference range.

C. Has undergone irreversible sterilization, including hysterectomy, bilateral oophorectomy or bilateral salpingectomy, except for bilateral tubal ligation.

8. Male patients should use barrier contraception (i.e., condoms) from screening until 3 months after treatment is discontinued.

9. The subject is willing to participate and sign the informed consent in person.

Exclusion Criteria:

* 1. Received any of the following treatments: A. Patients had undergone major surgery within 4 weeks before the first administration of the study drug; B. Received more than 30% of bone marrow irradiation or extensive radiotherapy within 4 weeks before the first administration of the drug; C. Within 7 days before the first administration of the study drug, CYP3A4 inhibitory agent, inducer or drug with narrow therapeutic window for CYP3A4 sensitive substrate was used.

  2. Patients with other malignancies requiring standard treatment or major surgery within 2 years of the first administration of the treatment under study.

  3. At the time of initiation of treatment, there was residual toxicity from previous treatment that was not alleviated, greater than CTCAE level 1, except for hair loss and level 2 neurotoxicity caused by previous chemotherapy.

  4. Spinal cord compression or brain metastases, unless asymptomatic, stable, and not requiring steroid therapy at least 2 weeks prior to the first administration of the study treatment.

  5. At the investigator's discretion, there were any serious or poorly controlled systemic diseases, such as poorly controlled hypertension, active bleeding constitutions, or active infections. There is no need to screen for chronic diseases.

  6. Refractory nausea, vomiting, or chronic gastrointestinal disease, inability to swallow research drugs, or a history of extensive bowel resection, may interfere with adequate absorption of amitinib.

  7. Meet any of the following cardiac examination results: A. mean correction of QT interval (QTc) > 470 msec obtained by 3 electrocardiogram (ECG) examinations in resting state, and QT interval correction (QTcF) was performed using Fridericia formula; B. The resting ECG indicated a variety of clinically significant rhythms and morphological abnormalities in the conduction or ECG (such as complete left bundle branch block, degree 3 atrioventricular block, degree 2 atrioventricular block, and PR interval > 250 msec).

C. Presence of any factor that increases the risk of prolonged QTc or arrhythmia events, such as heart failure, hypokalemia, congenital long QT syndrome, a family history of long QT syndrome, or sudden unexplained death in immediate family members under 40 years of age, or any combination of medications that prolong the QT interval; D. Left ventricular ejection fraction (LVEF) ≤40%. 8. A history of interstitial lung disease, a history of drug-induced interstitial lung disease, a history of radiation pneumonia requiring steroid treatment, or any evidence of clinically active interstitial lung disease.

9. Insufficient bone marrow reserve or organ function to achieve the following laboratory limits: A. Absolute neutrophil count <1.5×109 / L; B. Platelet count <100×109 / L; C. Hemoglobin <90 g/L (<9 g/dL); D. If there is no clear liver metastasis, the upper limit (ULN) of alanine aminotransferase > is 2.5 times normal; If there is liver metastasis, alanine aminotransferase > 5×ULN; E. If there is no definite liver metastasis, aspartate aminotransferase > 2.5×ULN; If there is liver metastasis, aspartic acid aminotransferase > 5×ULN; F. If there is no definite liver metastasis, total bilirubin > 1.5×ULN; Gilbert syndrome (unbound hyperbilirubinemia) or liver metastasis, total bilirubin > 3×ULN; G. Creatinine > 1.5×ULN and creatinine clearance <50 mL/min (calculated by Cockcroft - Gault formula); Confirmation of creatinine clearance is required only if creatinine > 1.5×ULN.

10. Women during lactation or in the study who had positive blood or urine pregnancy test results within 3 days before the first administration of treatment.

11. A history of hypersensitivity to any active or inactive component of amitinib or to drugs chemically similar to or similar to amitinib.

12. A history of hypersensitivity to any active or inactive component of pyrrolitinib or to drugs chemically similar to or similar to pyrrolitinib.

13. Any serious or uncontrolled ocular lesions that may, in the judgment of the physician, increase the patient's safety risk.

14. Patients identified by the investigator as likely to have poor compliance with study procedures and requirements.

15. Patients identified by the investigator as having any condition that jeopardizes patient safety or interferes with study evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 36 months
  Security of Almonertinib combined with Pyrotinib in the treatment of advanced NSCLC patients with HER-2 amplification/mutation after EGFR-TKI resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No